CLINICAL TRIAL: NCT02402608
Title: Whey Protein, Amino Acids and Vitamin D Supplementation With Physical Activity Increases Muscle Mass and Strength, Functionality and Quality of Life and Decreases Inflammation in Sarcopenic Elderly
Brief Title: Efficacy of Dietary Supplementation and Physical Activity in Sarcopenic Elderly
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda di Servizi alla Persona di Pavia (Other)
Collaborators: University of Pavia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: ASP-1
Record Dates: First submitted 2015-03-22; First posted 2015-03-30 (Estimated); Last update posted 2015-03-30 (Estimated); Status verified 2015-03

CONDITIONS: Sarcopenia
MeSH Terms: conditions — Sarcopenia | interventions — Dietary Supplements

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- dietary supplement (Active Comparator): oral essential amino acid (EAA), whey protein and vitamin D mixture (32 g)
  Interventions: Dietary Supplement: dietary supplement
- placebo (Placebo Comparator): placebo consisting of an equicaloric amount of maltodextrin with the same flavour and appearance as for the intervention product
  Interventions: Dietary Supplement: placebo

INTERVENTIONS:
Dietary Supplement: dietary supplement — oral essential amino acid (EAA), whey protein and vitamin D mixture
  Arms: dietary supplement
Dietary Supplement: placebo — placebo consisting of an equicaloric amount of maltodextrin with the same flavour and appearance as for the intervention product
  Arms: placebo

SUMMARY:
This 3 months randomized, double-blind, placebo-controlled supplementation trial tested the hypothesis that nutritional supplementation with whey protein, essential amino acids and vitamin D concurrent with regular, controlled physical activity would increase muscle mass, strength, physical functional, quality of life, and decrease the risk of malnutrition and inflammation in sarcopenic elderly.

DETAILED DESCRIPTION:
This 3 months randomized, double-blind, placebo-controlled supplementation trial tested the hypothesis that nutritional supplementation (32 g) with whey protein, essential amino acids and vitamin D concurrent with regular, controlled physical activity would increase muscle mass (assessed by DXA), strength (assessed by handgrip dynamometer), physical functional (assessed by ADL), quality of life (assessed by SF-36), and decrease the risk of malnutrition (assessed by MNA and IGF-I) and inflammation (assessed by C-reactive protein) in sarcopenic elderly.

ELIGIBILITY:
Inclusion Criteria:

* Eligible patients were aged 65 years or older with appendicular skeletal muscle mass/height2 2SD below mean of young adults (Baumgartner R, 1998), so with relative muscle mass < 7.26 kg/m2 for men and < 5.5 kg/m2 for women.
* Patients were not affected by acute illness, severe liver, heart or kidney dysfunction, and had a body weight which had been stable for 6 months

Exclusion Criteria:

* Subjects with altered glycometabolic control, disthyroidism and other endocrinopathies and cancers, as well as patients treated with steroids and heparin, or with total walking incapacity were excluded.

Ages: 65 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 130 (Actual)
Dates: Start 2012-01; Primary Completion 2014-11 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
muscle mass assessed by dual x-ray absorptiometry | 3 months
  muscle mass assessed by dual x-ray absorptiometry

SECONDARY OUTCOMES:
muscle strength assessed by handgrip dynamometer | 3 months
  muscle strength assessed by handgrip dynamometer
quality of life assessed by SF-36 | 3 months
  quality of life assessed by SF-36
inflammation assessed by C-reactive protein | 3 months
  inflammation assessed by C-reactive protein
malnutrition assessed by Mini Nutritional Assessment | 3 months
  malnutrition assessed by Mini Nutritional Assessment
functionality assessed by activity daily living | 3 months
  assessed by activity daily living
fat mass distribution assessed by DXA | 3 months
  body composition assessed by DXA
GH-IGF-I axsis by Insulin like growth factor -I (IGF-I) | 3 months
  Insulin like growth factor -I (IGF-I)

CONTACTS AND LOCATIONS:
Overall Officials: mariangela rondanelli, MD, PhD, Principal Investigator — University of Pavia
Locations (1):
- geriatric physical medicine and rehabilitation division at the Istituto Santa Margherita, Azienda di Servizi alla Persona di Pavia, Pavia, Pavia, Italy

REFERENCES:
- [Background] Rondanelli M, Faliva M, Monteferrario F, Peroni G, Repaci E, Allieri F, Perna S. Novel insights on nutrient management of sarcopenia in elderly. Biomed Res Int. 2015;2015:524948. doi: 10.1155/2015/524948. Epub 2015 Jan 29. PMID 25705670
- [Background] Bjorkman MP, Suominen MH, Pitkala KH, Finne-Soveri HU, Tilvis RS. Porvoo sarcopenia and nutrition trial: effects of protein supplementation on functional performance in home-dwelling sarcopenic older people - study protocol for a randomized controlled trial. Trials. 2013 Nov 14;14:387. doi: 10.1186/1745-6215-14-387. PMID 24225081
- [Derived] Rondanelli M, Klersy C, Terracol G, Talluri J, Maugeri R, Guido D, Faliva MA, Solerte BS, Fioravanti M, Lukaski H, Perna S. Whey protein, amino acids, and vitamin D supplementation with physical activity increases fat-free mass and strength, functionality, and quality of life and decreases inflammation in sarcopenic elderly. Am J Clin Nutr. 2016 Mar;103(3):830-40. doi: 10.3945/ajcn.115.113357. Epub 2016 Feb 10. PMID 26864356